CLINICAL TRIAL: NCT02312622
Title: A Phase 2 Study of Etirinotecan Pegol (NKTR-102) in Patients With Refractory Brain Metastases and Advanced Lung Cancer or Metastatic Breast Cancer (MBC)
Brief Title: Phase 2 Etirinotecan Pegol in Refractory Brain Metastases & Advanced Lung Cancer / Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joel Neal (Other)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Joel Neal, ASSISTANT PROFESSOR OF MEDICINE, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-30982; NCI-2014-02101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LUN0067 (Other: OnCore); IRB-30982 (Other: Stanford University IRB)
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Stage IV Non-small Cell Lung Cancer (NSCLC); Recurrent Non-small Cell Lung Cancer (NSCLC); Extensive-stage Small Cell Lung Cancer (SCLC); Recurrent Small Cell Lung Cancer (SCLC); Tumors Metastatic to Brain; Metastatic Breast Cancer (mBC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Brain Neoplasms; Breast Neoplasms | interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A - Pegylated Irinotecan to treat NSCLC (Experimental): Patients with non-small cell lung carinoma (NSCLC) will receive pegylated irinotecan intravenously (IV) over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pegylated Irinotecan
- Cohort B - Pegylated Irinotecan to treat SCLC (Experimental): Patients with small cell lung carinoma (SCLC) will receive pegylated irinotecan intravenously (IV) over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pegylated Irinotecan
- Cohort C - Pegylated Irinotecan to treat mBC (Experimental): Patients with metastatic breast cancer (MBC) to brain will receive pegylated irinotecan intravenously (IV) over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pegylated Irinotecan

INTERVENTIONS:
Drug: Pegylated Irinotecan — Administered intravenously (IV) at 145 mg/m² as monotherapy once every 21 days (1 cycle)
  Other Names: NKTR-102; PEG-irinotecan; etirinotecan pegol

SUMMARY:
This phase 2 trial evaluates how well pegylated irinotecan (NKTR-102) works in treating patients with non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC), or breast cancer (mBC) that has spread to the brain and does not respond to treatment. Pegylated irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
Primary Objective:

For cohort A and Cohort C, to determine the central nervous system (CNS) disease control rate (number of patients with stable disease or partial response or complete response / total number of treated patients) at 12 weeks following treatment with etirinotecan pegol in patients with advanced non-small cell lung cancer (NSCLC) or with metastatic brain cancer (mBC) with refractory brain metastases

Secondary Objectives:

Cohorts A and C:

* To measure the overall disease control rate and response rate for patients receiving study therapy
* To measure the systemic (non-CNS) disease control rate and response rate for patients receiving study therapy
* To observe the progression free survival of the study population
* To observe the overall survival of the study population

Cohort B:

• To observe CNS and systemic disease control in small cell lung cancer (SCLC)

Cohorts A, B and C:

• To determine the safety profile of etirinotecan pegol

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Life expectancy of 3 months or longer.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Advanced or refractory cancer, consisting of

* Metastatic breast cancer (mBC) for which single-agent cytotoxic chemotherapy is indicated. OR
* Histologically-proven metastatic lung cancer:

  * Non-small cell lung cancer (NSCLC) as Stage IV disease or recurrent metastatic disease [per lung cancer tumor, node and metastasis (TNM) classification system, 7th ed] (Cohort A) OR
  * Small cell lung cancer (SCLC) as extensive stage or recurrent metastatic disease (cohort B), including tumors with mixed small cell and non-small cell elements.

Prior chemotherapy (at least one of the following):

* At least one line of prior systemic chemotherapy
* At least one line of prior targeted treatment for metastatic disease Adjuvant systemic chemotherapy within prior 6 months Prior treatment for metastatic breast cancer (mBC) must have included taxane-based regimen

Prior chemotherapy, including other investigational therapy, has been completed prior to initiation of study treatment, according to the following:

* ≥ 2 weeks if immediately preceding treatment was chemotherapy/targeted therapy administered on a daily or weekly schedule
* ≥ 3 weeks if immediately preceding treatment was chemotherapy/targeted therapy administered every 2 weeks
* ≥ 4 weeks if immediately preceding treatment was chemotherapy/targeted therapy administered every 3 weeks Previously received at least one CNS directed treatment (such as surgery or radiation) OR not be eligible for CNS stereotactic radiosurgery Measurable CNS disease, either previously untreated (not counting systemic therapy), or progressed following previous radiation treatment. Lesions that have progressed after prior radiosurgery should not be selected as measurable disease if they are suspected of being radionecrosis.

The following measurement criteria are required, as visualized by contrast-enhanced MRI with slice thickness of ≤ 1.5 mm, unless absence of contrast or thicker slices is specifically authorized by Protocol Director. Measurements do not include tumor edema.

* At least one CNS tumor measuring ≥ 10 mm in longest diameter, OR
* At least one CNS tumor measuring 5-9 mm in longest diameter, plus one or two additional CNS tumors measuring ≥ 3 mm in longest diameter, for which the sum of the longest diameters is ≥ 10 mm. Additional tumors are not exclusionary.

Adequate organ function as evidenced by:

* Absolute neutrophil count (ANC) ≥ 1.5 x 10e9/L without G-CSF (filgrastim, pegfilgrastim, or equivalent) support within 7 days
* Hemoglobin (Hgb) ≥ 9.0 g/dL (90 g/L) without blood transfusion within 7 days
* Platelet count ≥ 100 x 10e9/L without platelet transfusion within 7 days
* Bilirubin ≤ 1.5 X upper limit of normal (ULN), except for patients with documented history of Gilbert's disease who may have DIRECT bilirubin ≤ 1.5 X ULN
* Alanine aminotransferase (ALT) ≤ 2.5 X ULN, except ≤ 5 X ULN for patients with liver metastases
* Aspartate aminotransferase (AST) ≤ 2.5 X ULN, except ≤ 5 X ULN for patients with liver metastases
* Serum creatinine ≤ 1.5 X ULN; or calculated creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula), or measured creatinine clearance ≥ 50 mL/min.

Exclusion Criteria:

* Previous treatment with a camptothecin derivative (eg, irinotecan, topotecan, and investigational agents including but not limited to exatecan, rubitecan, gimatecan, karenitecin, SN38 investigational agents, EZN 2208, SN 2310, and AR 67) is not allowed
* Patients may not have a known history of leptomeningeal disease, as diagnosed by positive CSF cytology, unless prospective permission for enrollment is granted from the sponsor and the PI
* Patients may not have had major surgery or radiotherapy (therapeutic and/or palliative) within 14 days prior to initiation of study treatment, including CNS-directed radiation therapy. Minor procedures, such as tumor biopsy, thoracentesis, or intravenous catheter placement are allowed with no waiting period
* Patients may not have the following co morbid disease or concurrent illness:

  * Chronic or acute gastrointestinal (GI) disorders resulting in diarrhea of any severity grade; patients may not use chronic anti-diarrheal supportive care (more than 3 days/week) to control diarrhea in the 28 days prior to first dose of investigational drug. (exception: anti-diarrheal medications used to control symptoms from a medication that will be discontinued prior to study are allowed with a 7 day washout before study therapy, for example loperamide for erlotinib-associated diarrhea)
  * Known cirrhosis, defined as Child Pugh class A or higher liver disease
  * Other active malignancy, except for non melanoma skin cancer and carcinoma in situ (of the cervix or bladder)
  * Any other severe/uncontrolled inter current illness or significant co morbid conditions that in the opinion of the investigator would impair study participation or cooperation
* Patients may not have a known allergy or hypersensitivity to any of the components of the investigational therapy, including polyethylene glycol (PEG) or topoisomerase inhibitors
* Patients may not be receiving the following medications at the time of first dose of investigational drug:

  * Pharmacotherapy for known hepatitis B or C, tuberculosis, or human immunodeficiency virus (HIV)
  * Any of the following enzyme inducing anti epileptic medications (EIAEDs): phenytoin, carbamazepine, oxcarbazepine, phenobarbital
  * Other chemotherapy, hormonal therapy, immunotherapy, other investigational agents, or biologic agents for the treatment of cancer except for bisphosphonates or denosumab
* Pregnant or nursing patients will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-08; Primary Completion 2018-09-08 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neal, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A - Pegylated Irinotecan to Treat NSCLC: Patients with non-small cell lung carinoma (NSCLC) will receive pegylated irinotecan NKTR 102 IV over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Pegylated Irinotecan: Administered intravenously (IV) at 145 mg/m² as monotherapy once every 21 days (1 cycle)
- Cohort B - Pegylated Irinotecan to Treat SCLC: Patients with small cell lung carinoma (SCLC) will receive pegylated irinotecan NKTR 102 IV over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Pegylated Irinotecan: Administered intravenously (IV) at 145 mg/m² as monotherapy once every 21 days (1 cycle)
- Cohort C - Pegylated Irinotecan to Treat mBC: Patients with metastatic breast cancer (MBC) to brain will receive pegylated irinotecan NKTR 102 IV over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Pegylated Irinotecan: Administered intravenously (IV) at 145 mg/m² as monotherapy once every 21 days (1 cycle)
Period: Overall Study
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort B - Pegylated Irinotecan to Treat SCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Started | 12 | 3 | 12
Completed | 12 | 3 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort B - Pegylated Irinotecan to Treat SCLC | Cohort C - Pegylated Irinotecan to Treat mBC | Total
Number analyzed (Participants) | 12 | 3 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 2 | 11 | 22
  >=65 years | 3 | 1 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.2) | 63.3 (15.5) | 48.2 (10.9) | 53.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 12 | 22
  Male | 4 | 1 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 3 | 11 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 0 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 10 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Disease Control Rate (Cohort A and C)
Description: Central nervous system (CNS) disease control (DC) is defined as a complete response (CR); partial response (PR); or stable disease (SD). The outcome is reported as the number and percentage of participants who achieve DC, a number without dispersion.
  Response criteria are as follows. Note that any lesion less than 10 mm in longest diameter (LD) is considered unchanged unless there is a ≥ 3 mm change in the sum of the LDs.
  * CR = Disappearance of all target lesions, sustained for ≥ 4 weeks with no new lesions; clinical condition stable or improved
  * PR = ≥ 30% decrease in target lesion LD and no new lesions, sustained for ≥ 4 weeks; clinical condition stable or improved
  * PD (progressive disease) = Any of 20% increase in target lesion LD; increase in T2/FLAIR non-enhancing lesions; any new lesions; non-target progression; or clinical deterioration
  * SD = Neither PR or PD
Time Frame: At 12 weeks
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
Participants | 2 | 2

2. Secondary Outcome: Overall Disease Control Rate (Cohort A and C)
Description: Overall disease control (DC) rate is defined as the sum in a cohort of the numbers of participants achieving complete response (CR); partial response (PR); or stable disease (SD), divided by the number of patients in that cohort. For this outcome, "overall" means all body systems, not just the central nervous system (CNS). The outcome is reported as DC rate, a number without dispersion.
  Response criteria are as follows. Note that any lesion <10 mm in longest diameter (LD) is considered unchanged unless there is a ≥3 mm change in the sum of the LDs.
  * CR = Disappearance of all target lesions, sustained for ≥4 weeks with no new lesions; clinical condition stable or improved
  * PR = ≥30% decrease in target lesion LD & no new lesions, sustained for ≥ 4 weeks; clinical condition stable or improved
  * PD = Any of: 20% increase in target lesion LD; increase in T2/FLAIR non-enhancing lesions; any new lesions; non-target progression; or clinical deterioration
  * SD = Neither PR or PD
Time Frame: At 12 weeks
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Number; unit: participants
Groups:
- Cohort C - Pegylated Irinotecan to Treat mBC: Cohort C - Pegylated Irinotecan to treat mBC Patients with metastatic breast cancer (MBC) to brain will receive pegylated irinotecan intravenously (IV) over 90 minutes every 21 days in the absence of disease progression or unacceptable toxicity.
  Pegylated Irinotecan: Administered intravenously (IV) at 145 mg/m² as monotherapy once every 21 days (1 cycle)
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
participants | 2 | 2

3. Secondary Outcome: Overall Response Rate (Cohort A and C)
Description: Overall response by subject (OR) is defined as the lower assessment between the central nervous system response and the systemic response. Response is defined as either complete response (CR) or partial response (PR). The outcome is reported as the number and percentage of participants who achieve OR, a number without dispersion.
  Response criteria are as follows. Note that any lesion < 10 mm in longest diameter (LD) is considered unchanged unless there is a ≥ 3 mm change in the sum of the LDs.
  * CR = Disappearance of all lesions, sustained for ≥ 4 weeks with no new lesions; clinical condition stable or improved
  * PR = ≥ 30% decrease in target lesion LD & no new lesions, sustained for ≥ 4 weeks; clinical condition stable or improved
  * PD = Any of: 20% increase in target lesion LD; increase in T2/FLAIR non-enhancing lesions; any new lesions; non-target progression; or clinical deterioration
  * SD = Neither PR or PD
Time Frame: At 12 weeks
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
Participants | 1 | 0

4. Secondary Outcome: Systemic (Non-CNS) Disease Control Rate (Cohort A and C)
Description: Systemic (ie, non-central nervous system) disease control (DC) rate by cohort is defined as the number of patients with complete response (CR) + partial response (PR) + stable disease (SD), divided by the total number of patients. The outcome will be reported as DC rate, a number without dispersion.
  Response criteria are as follows. Note that any lesion < 10 mm in longest diameter (LD) is considered unchanged unless there is a ≥ 3 mm change in the sum of the LDs.
  * CR = Disappearance of all lesions, no new lesions; pathological lymph nodes reduced in short axis to < 10 mm
  * PR = ≥ 30% decrease in sum of lesion diameters; no new lesions; no progression of non-target lesions
  * PD = Any of 20% increase in sum of lesion diameters; progression of non-target lesions; new lesions
  * SD = Neither CR, PR, nor PD
Time Frame: At 12 weeks
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
Participants | 3 | 3

5. Secondary Outcome: Systemic (Non-CNS) Response Rate (Cohort A and C)
Description: Systemic (ie, non-central nervous system) response rate by cohort is defined as the number of participants achieving a complete response (CR) or partial response (PR), divided by the number of participants. The outcome will be reported as a number without dispersion.
  Response criteria are as follows. Note that any lesion < 10 mm in longest diameter (LD) is considered unchanged unless there is a ≥ 3 mm change in the sum of the LDs.
  * CR = Disappearance of all target lesions, no new lesions; pathological lymph nodes reduced in short axis to < 10 mm
  * PR = ≥ 30% decrease in sum of lesion diameters; no new lesions; no progression of non-target lesions
  * PD = Any of 20% increase in sum of lesion diameters; progression of non-target lesions; new lesions
  * SD = Neither CR, PR, nor PD
Time Frame: At 12 weeks
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
Participants | 1 | 0

6. Secondary Outcome: Progression-free Survival (PFS) (Cohort A and C)
Description: Progression-free survival (PFS) is defined as the time from the date of start of treatment until disease progression or death. The outcome is reported by cohort as PFS in months, with full range.
Time Frame: Date of first dose of pegylated irinotecan NKTR 102 to date of disease progression, assessed up to 2 years
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
months | 2.66 [1.35 to 6.74] | 1.35 [1.31 to 6.88]

7. Secondary Outcome: Overall Survival (Cohort A and C)
Description: Overall survival (OS) is defined as the period remaining alive after the start of treatment. The outcome is reported as the median with full range.
Time Frame: 4 years
Population: Cohort B (metastatic small cell lung cancer, SCLC) is excluded per protocol from this outcome.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 12
months | 7.00 [5.13 to 48] | 8.49 [1.94 to 21.84]

8. Secondary Outcome: Central Nervous System (CNS) Disease Control (Cohort B)
Description: Central nervous system (CNS) disease control (DC) is defined as a complete response (CR); partial response (PR); or stable disease (SD). The outcome is reported as the number and percentage of participants who achieve DC, a number without dispersion.
  Response criteria are as follows. Note that any lesion less than 10 mm in longest diameter (LD) is considered unchanged unless there is a ≥ 3 mm change in the sum of the LDs.
  * CR = Disappearance of all target lesions, sustained for ≥ 4 weeks with no new lesions; clinical condition stable or improved
  * PR = ≥ 30% decrease in target lesion LD and no new lesions, sustained for ≥ 4 weeks; clinical condition stable or improved
  * PD = Any of 20% increase in target lesion LD; increase in T2/FLAIR non-enhancing lesions; any new lesions; non-target progression; or clinical deterioration
  * SD = Neither PR or PD
Time Frame: At 12 weeks
Population: This outcome was restricted by protocol to Cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B - Pegylated Irinotecan to Treat SCLC
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Systemic Disease Control (Cohort B)
Description: as for outcome 4
Time Frame: At 12 weeks
Population: This outcome was restricted by protocol to Cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B - Pegylated Irinotecan to Treat SCLC
Number analyzed (Participants) | 3
Participants | 0

10. Secondary Outcome: Related Adverse Events (Toxicity)
Description: Toxicity, defined as related adverse events, is reported as the total number of events experienced by the participants in each cohort, a number without dispersion. Related is defined as meaning possibly, probably, or definitely related to the study drug.
Time Frame: Up to 2 years
Population: All participants are included.
Measure: Number; unit: adverse events
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort B - Pegylated Irinotecan to Treat SCLC | Cohort C - Pegylated Irinotecan to Treat mBC
Number analyzed (Participants) | 12 | 3 | 12
adverse events | 70 | 40 | 68

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort A - Pegylated Irinotecan to Treat NSCLC | Cohort B - Pegylated Irinotecan to Treat SCLC | Cohort C - Pegylated Irinotecan to Treat mBC
All-Cause Mortality (participants affected / at risk) | 11/12 | 3/3 | 11/12
Serious Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 6/12
Other Adverse Events (participants affected / at risk) | 12/12 | 3/3 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Pegylated Irinotecan to Treat NSCLC (N=12) | Cohort B - Pegylated Irinotecan to Treat SCLC (N=3) | Cohort C - Pegylated Irinotecan to Treat mBC (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Pegylated Irinotecan to Treat NSCLC (N=12) | Cohort B - Pegylated Irinotecan to Treat SCLC (N=3) | Cohort C - Pegylated Irinotecan to Treat mBC (N=12)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (3)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Anal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 3 (4) | 1 (2) | 2 (2)
Body Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (26) | 3 (9) | 5 (25)
Double vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Edema Face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (5) | 5 (7)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (4) | 0 (0) | 3 (4)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion Related reaction (General disorders) | 1 (2) | 0 (0) | 1 (2)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (13) | 2 (4) | 4 (6)
Non Cardiac Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oral Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 3 (4) | 1 (2) | 1 (1)
Pupil Constriction (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Right Eye Redness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (14) | 1 (1) | 3 (4)
Weight Loss (Investigations) | 1 (1) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
White Blood Cell Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Multifocal Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mild Transaminitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Vaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 2 (4) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular Menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (2) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash manuco-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Shock Liver (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT02312622/Prot_SAP_000.pdf